CLINICAL TRIAL: NCT06348329
Title: The Effect of Pregnant Women Participating in Birth Preparation Training With Their Spouses on the Parenting Role, Attitudes of Their Spouses Towards Participating in the Birth, and Birth Self-Efficacy
Brief Title: Pregnant Women Participating in Birth Preparation Training With Their Spouses on the Parenting Role, Attitudes of Their Spouses Towards Participating in the Birth, and Birth Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Principal Investigator, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TÜTF-GOBAEK 2023/41
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Birth Order; Parenting; Self Efficacy; Pregnancy Related
Keywords: Birth Preparation Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education without co-participation (Experimental)
  Interventions: Other: Birth Preparation Training
- education with co-participation (Experimental)
  Interventions: Other: Birth Preparation Training

INTERVENTIONS:
Other: Birth Preparation Training — Birth Preparation Training is planned to include a 4-week program by an internationally certified instructor.

SUMMARY:
In this prospective, randomized controlled study, it was aimed to examine the effect of pregnant women participating in birth preparation training together with their partners on the parenting role, spouses' attitudes towards participation in birth, and birth self-efficacy.

The study was shared via the web on social media (Facebook, Instagram, Twitter, Telegram) forum pages between 25.09.2023-25.03.2025, and n=158 pregnant women who met the inclusion criteria and volunteered to participate in the study (79= education without spouse participation, 79= spouse Participatory education) will be conducted randomly in two groups: case and control.

Before starting the research, two groups will be randomly formed among pregnant women. As a randomization method, pregnant women who meet the sampling inclusion criteria determined in the research will be identified and listed. Individuals to be taken into two groups will be determined by randomization method from the random numbers table. (http://www.stattrek.com/statistics/randomnumber-generator.aspx).

DETAILED DESCRIPTION:
The study was shared via the web on social media (Facebook, Instagram, Twitter, Telegram) forum pages between 25.09.2023-25.03.2025, and n=158 pregnant women who met the inclusion criteria and volunteered to participate in the study (79= education without spouse participation, 79= spouse Participatory education) will be conducted randomly in two groups: case and control.

Since the study is descriptive in nature, it was calculated that 158 pregnant women should be included in the study in order to determine the scale score regarding the "Spouse Support Scale" score with an 80% effect level, 95% confidence level and 5% margin of error.

Before starting the research, two groups will be randomly formed among pregnant women. As a randomization method, pregnant women who meet the sampling inclusion criteria determined in the research will be identified and listed. Individuals to be taken into two groups will be determined by randomization method from the random numbers table. (http://www.stattrek.com/statistics/randomnumber-generator.aspx).

In the first interview for both groups, "Information Form", "Postpartum Parenting Behavior Scale", "Self-Efficacy Scale in Labor", "Attitude Scale towards Participating in Birth for Expectant Fathers" and "Spouse Support Scale" were given to each participant with information about the study. After the purpose of the study is explained, an e-survey containing survey and scale questions will be used. The e-survey will be arranged so that each participant participates only once. In the first part of the e-survey, information about the study and the purpose of the study will be explained to the pregnant women, and if they confirm that they want to participate, they will begin the second part, the survey questions. Pregnant women assigned to the training group are included in the Birth Preparation Class and taught online for 4 weeks, once a week, for an average of 3 hours a day. They will be asked to participate in the ongoing training with their spouses. All scales will be repeated before training, after training and in the 1st month after birth. Birth Preparation Training will be provided by a certified educator and researcher who has training in the field.

In the study, the "Information Form", "Postpartum Parenting Behavior Scale", "Self-Efficacy in Labor Scale", "Attitude Scale towards Participating in Birth for Expectant Fathers" and "Spouse Support Scale" prepared by the researchers will be used.

Information Form: It was created by researchers by scanning the literature and consists of a total of 28 questions: 15 questions covering the socio-demographic characteristics of pregnant women, 7 questions covering their obstetric characteristics, and 6 questions about their thoughts on labor.

Postnatal Parenting Behavior Scale: It is used to evaluate the parenting behavior of parents towards the baby during their first encounter with their baby after birth. The scale can only be applied to parents in the first minutes after birth. The scale, which consists of items such as close contact, touching with affection, examining the baby, talking with affection, positive comments and happiness, is evaluated in a binary scoring manner by marking these items as present/absent. Each item is evaluated as one (1) point if the behavior is observed, and zero (0) point if the behavior is not observed. The total scale score consists of the sum of the numbers obtained from each item. The total score of the scale is between 0-6 points. A higher total score from the scale indicates that the parent has more positive parenting behavior towards his/her baby.

Self-Efficacy in Labor Scale: The Turkish validity and reliability study of the scale, which measures women's self-confidence and coing ability regarding labor, was conducted. The scale has two sub-dimensions: outcome and competence expectation. Each sub-dimension of the scale consists of 16 questions. The lowest score to be obtained from the scale sub-dimensions is 16 and the highest score is 160. High scores from the subscales indicate that pregnant women have high expectations of adequacy and outcome regarding birth. Responses on a Likert-type scale are scored from 1 to 10. In the outcome expectation sub-dimension of the scale; 1 is "not useful at all", 10 is "very useful", and in the proficiency expectation sub-dimension; The first 13 questions are marked as 1 "completely sure", 10 as "not at all sure", questions 14-16 as 1 "not at all sure", and 10 as "completely sure". Questions 1 to 13 in the proficiency expectation sub-dimension of the scale were scored in reverse order. The lowest total score that can be obtained from the scale is 32, and the highest total score is 320. High scores from the scale indicate that pregnant women have high self-efficacy levels in labor. Cronbach's alpha coefficient of the scale was found to be 0.90.

Spouse Support Scale: The scale developed is used to measure the support spouses receive from each other. The scale consists of a total of 27 questions, and there are 3 reversed items. The scale has a three-point rating; It is shown as Suitable for Me=3, Partially Suitable for Me=2, Not Suitable for Me=1. Just like straight items, reversed items are scored in reverse. The scale has four factors. The first factor is 'emotional support' (6,16,12,21,4,1,3,9,2) consisting of nine items, and the second factor is 'financial aid and information support' (24,17,27,25,13,7, 15) consists of seven items, the third factor 'appreciation support' (18,10,5,26,14,22,23,20) consists of eight items, and the fourth factor 'social interest support' (19,11,8) consists of three items. The score that can be obtained from EDS varies between 27-81. The lower the score, the less support, the higher the score, the more support. The Cronbach Alpha coefficient of the scale is stated as 0.95.

Attitude Scale for Father Candidates Towards Participating in the Birth: The scale is used to evaluate the attitudes of father candidates towards attending the birth. The scale consists of 26 items and is a five-point Likert type. The reactions of the prospective fathers who answered the scale to the items are measured with five options for positive statements, depending on their degree of agreement: completely agree = 5, agree = 4, undecided = 3, disagree = 2, completely disagree = 1. The scale contains 18 positive items and 8 negative items. Negative expressions are coded by reversing. The scale consists of three subscales: Positive Emotions Towards Participating in Birth, Negative Emotions Towards Participating in Birth, and Actions Towards Participating in Birth. The lowest score that can be obtained from the scale is 26 and the highest score is 130. An increase in the total score of the scale indicates that prospective fathers have a more positive attitude towards participating in the birth. The decrease in the total score shows that prospective fathers have a negative attitude towards participating in the birth.

ELIGIBILITY:
Inclusion Criteria:

• Over the age of 18, the mother and the baby must not have any health problems during pregnancy, birth and postpartum period, do not have a previously diagnosed mental disorder, must attend the Birth Preparation Class (BPC) with their spouses for the group receiving co-participation training and continue for 4 weeks. For the education group without partner participation, pregnant women who do not participate in the Birth Preparation Class (BPC) with their partners and continue for 4 weeks and who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

• Under the age of 18, having a health problem in the mother and the baby during pregnancy, birth and postpartum period, having a previously diagnosed mental disorder, not participating in the Birth Preparation Class (BPC) with their spouses for the group receiving training with partner participation and not attending the Birth Preparation Class (DHS) for 4 weeks. For the training group without partner participation, participation in the Birth Preparation Class (BPC) with their spouses and non-attendance for 4 weeks, and non-pregnant women will not be included in the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Parenting behavior evaluated using the Postpartum Parenting Behavior Scale | change from baseline implamentation patent and after training and 1st month after birth of practice
  It is used to evaluate the parenting behavior of parents towards the baby during their first encounter with their baby after birth. The scale can only be applied to parents in the first minutes after birth. Britton et al. It was developed by Çalışır et al. Turkish validity and reliability were conducted by. The scale, which consists of items such as close contact, touching with affection, examining the baby, talking with affection, positive comments and happiness, is evaluated in a binary scoring manner by marking these items as present/absent. Each item is evaluated as one (1) point if the behavior is observed, and zero (0) point if the behavior is not observed. The total scale score consists of the sum of the numbers obtained from each item. The total score of the scale is between 0-6 points. A higher total score from the scale indicates that the parent has more positive parenting behavior towards his/her baby.
Parenting self-efficacy in labor evaluated using the Self-Efficacy in Labor Scale | change from baseline implamentation patent and after training and 1st month after birth of practice
  he Turkish validity and reliability study of the scale, which measures women's self-confidence and coping ability regarding labor, was conducted by Ersoy. The scale has two sub-dimensions: outcome and competence expectation. Each sub-dimension of the scale consists of 16 questions. The lowest score to be obtained from the scale sub-dimensions is 16 and the highest score is 160. High scores from the subscales indicate that pregnant women have high expectations of adequacy and outcome regarding birth. Responses on a Likert-type scale are scored from 1 to 10.
Spouse support evaluated using the Spouse Support Scale | change from baseline implamentation patent and after training and 1st month after birth of practice
  The scale developed by Yıldırım (2004) is used to measure the support spouses receive from each other. The scale consists of a total of 27 questions, and there are 3 reversed items (10,20,24). The scale has a three-point rating; It is shown as Suitable for Me=3, Partially Suitable for Me=2, Not Suitable for Me=1. Just like straight items, reversed items are scored in reverse. The scale has four factors. The first factor is 'emotional support' (6,16,12,21,4,1,3,9,2) consisting of nine items, and the second factor is 'financial aid and information support' (24,17,27,25,13,7, 15) consists of seven items, the third factor 'appreciation support' (18,10,5,26,14,22,23,20) consists of eight items, and the fourth factor 'social interest support' (19,11,8) consists of three items. The score that can be obtained from EDS varies between 27-81. The lower the score, the less support, the higher the score, the more support. The Cronbach Alpha coefficient of the scale is stated as 0.95.
Father candidates towards participating in the birth evaluated using the Attitude Scale for Father Candidates Towards Participating in the Birth | change from baseline implamentation patent and after training and 1st month after birth of practice
  The scale developed by Çiçek Özdemir and Kan in 2022 is used to evaluate the attitudes of father candidates towards attending the birth. The scale consists of 26 items and is a five-point Likert type. The reactions of the prospective fathers who answered the scale to the items are measured with five options for positive statements, depending on their degree of agreement: completely agree = 5, agree = 4, undecided = 3, disagree = 2, completely disagree = 1. The scale contains 18 positive items and 8 negative items. Negative expressions are coded by reversing. The scale consists of three subscales: Positive Emotions Towards Participating in Birth, Negative Emotions Towards Participating in Birth, and Actions Towards Participating in Birth.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)